CLINICAL TRIAL: NCT07107997
Title: Transcranial Doppler Versus Computed Tomography In Evaluation Of Brain Edema In Patients With Traumatic Brain Injury
Brief Title: Transcranial Doppler in Traumatic Brain Edema
Acronym: TCD TBI
Status: Completed | Type: Observational
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Other Study IDs: 0108653
Record Dates: First submitted 2025-07-31; First posted 2025-08-06 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: Traumatic Brain Injury
Keywords: Transcranial Doppler; Traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Traumatic brain injury patients: Traumatic brain injury patients, with brain edema

SUMMARY:
The goal of this clinical trial is to assess the role of transcranial Doppler (TCD) in evaluating brain edema in traumatic brain injury. The main question it aims to answer is:

Is TCD equivalent to brain computerized tomography (CT) in evaluating traumatic brain edema?

Participants will be examined by both methods at the same time to assess the correlation between them.

DETAILED DESCRIPTION:
Computed Tomography (CT) scan of the brain will be done on admission to the ICU and 48-72 hours after starting hyperosmolar therapy. The cerebral oedema will be scored as follows: 0 = no brain oedema, 1 = mild brain oedema, 2 = moderate brain oedema, and 3 = severe brain oedema. Oedema is defined as mild when the ventricles and cisterns are narrow in the CT in the acute stage; moderate, when in addition to the mild form, the sylvian fissure and cortical gyri are not visualized; and severe, when in addition to mild and moderate, the perimesencephalic cisterns can not be visualized.

Transcranial doppler ultrasonography will be performed immediately after CT scan then after 48-72 hours of starting hyperosmolar therapy according to the following protocol:

* The examination will be done using phased array probe using (Versana active, general electric medical systems china Co.Ltd) ultrasound (US) device.
* Standing behind the head of the patient, the 2 Mega Hertz (MHz) transducer will be placed over the temporal area just above the zygomatic arch and in front of the tragus of the ear and oriented slightly upward and anteriorly.
* A red color signal (i.e. flow towards the probe) at a depth between 40-65 mm will represent the flow in the ipsilateral middle cerebral artery.
* The angle and position of insonation will be adjusted to provide the highest quality Doppler signal.
* By applying pulsed wave on the insonated segment, Peak Systolic Velocity (PSV) and End Diastolic Velocity (EDV) will be measured and recorded on US machine.
* Mean flow velocity (MFV) will be calculated using the formula:

(PSV+(EDVx 2))/3.

* Pulsatility index (PI) is calculated using the formula: (PSV-EDV)/ MFV.
* Intracranial pressure (ICP) will be calculated as follows:

  * CPP is calculated as: MAP*(EDV /MFV) + 14. where MAP is the mean arterial blood pressure.
  * ICP is then calculated as: MAP - CPP.

All patients in the study will be managed using the same management principles of traumatic brain injury with raised intracranial pressure such as:

* Hyperosmolar therapy either with 20% mannitol or 3% hypertonic saline.
* Control fever and seizures.
* Elevate head of bed 30-45.
* Adequate analgesia and sedation.
* Maintain systolic blood pressure > 90 mmHg.
* Maintain partial pressure of carbon dioxide (PaCo2) between 35-38 mmHg.
* Maintain partial pressure of oxygen (Pao2) between 80-120 mmHg.
* Avoid hyponatremia.
* Maintain Hb > 9 g/dL.

ELIGIBILITY:
Inclusion Criteria:

* Patients with brain edema following traumatic brain injury, admitted within 24 hours

Exclusion Criteria:

* Patients presented by out of hospital cardiac arrest or in-hospital cardiac arrest before performing the transcranial Doppler.
* Pregnant females.
* Inability to obtain adequate ultrasound window.
* Temporal bone fracture or brain herniation.
* Open head injuries or patients in need for surgical intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted to Critical Care Medicine Department in Alexandria University Hospitals
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2024-10-13 (Actual); Primary Completion 2025-04-13 (Actual); Study Completion 2025-06-13 (Actual)

PRIMARY OUTCOMES:
correlation between transcranial Doppler and brain CT in assessment of brain edema | 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Main University Hospital, Alexandria, Other (Specify), Egypt

IPD SHARING:
Plan to Share IPD: No